CLINICAL TRIAL: NCT03474458
Title: A Randomized Phase II/III Trial of Doxycycline vs. Standard Supportive Therapy in Newly-diagnosed Cardiac AL Amyloidosis Patients Undergoing Bortezomib-based Therapy
Brief Title: A Trial of Doxycycline vs. Standard Supportive Therapy in Newly-diagnosed Cardiac AL Amyloidosis Patients Undergoing Bortezomib-based Therapy
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: difficulty in recruitment
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Giovanni Palladini, Professor, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AC-012-EU
Record Dates: First submitted 2018-03-16; First posted 2018-03-22 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Cardiac AL Amyloidosis
MeSH Terms: interventions — Doxycycline

STUDY DESIGN:
Intervention Model Description: This will be an open-label parallel-group randomized (1:1) trial. Control patients receive standard supportive therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental intervention (Experimental): doxycycline (100 mg bid)
  Interventions: Drug: Doxycycline
- Control intervention (Active Comparator): Standard of care therapy
  Interventions: Drug: Standard of care therapy

INTERVENTIONS:
Drug: Doxycycline — Doxycycline
  Arms: Experimental intervention
Drug: Standard of care therapy — Standard of care therapy
  Arms: Control intervention

SUMMARY:
Systemic amyloidoses are rare diseases affecting approximately 1 in 100,000 persons each year.

In systemic amyloidoses abnormal proteins deposit in bodily organs and severely impair their function, causing death if not treated effectively. Light chain (AL) amyloidosis is caused by a usually small population of plasma cells (the cells that produce antibodies). These cells produce part of antibodies, the light chains (LC) that form amyloid deposits. Almost every organ, with the exception of the brain, can be affected by AL amyloidosis. The heart is involved in three fourths of patients and is responsible for almost all the deaths occurring in the first 6 months after diagnosis. Current therapy of AL amyloidosis is based on drugs targeting the plasma cells producing the amyloid-forming LC. At present, most patients receive a powerful anti-plasma cell drug, bortezomib, as part of their initial treatment. However, bortezomib-based therapy, can improve heart involvement only in less than one third of patients with AL amyloidosis, and many patients (approximately one third) still die within 12 months from diagnosis. Early cardiac deaths remain an acute unmet need and the major determinant of overall outcome in this disease. Thus, there is the need of alternative means to treat heart involvement in AL amyloidosis. Doxycycline is a widely used, well tolerated, antibiotic that has been marketed for decades and used to treat a number of different infectious diseases caused by bacteria. This molecule has been extensively studied in the laboratory, in animal models and, more recently, in small studies involving patients, for its potential of improving cardiac damage in amyloidosis. These studies showed that doxycycline disrupts amyloid deposits, reduces the amyloid load in a mouse model, and counteracts the toxicity exerted by amyloid-forming LCs on C. elegans, a worm whose pharynx is used as a model resembling human heart. In a small clinical study, doxycycline was given to patients with cardiac AL amyloidosis during treatment for their underlying plasma cell disease. This resulted in a remarkable improvement of survival compared to "matched historical controls" (i.e. similar patients who had received only anti-plasma cell therapy without doxycycline in the past). Based on these promising preliminary results, we designed the present clinical trial to assess whether the addition of doxycycline to anti-plasma cell therapy can improve survival in patients with cardiac AL amyloidosis who were not previously treated. The rate of survival at 12 months will be compared in patients receiving doxycycline and in controls receiving standard antibiotic therapy, together with anti-plasma cell therapy. Patients will be assessed for parameters of plasma cell disease, heart involvement and possible involvement of other organs, as well as for quality of life. To make sure that patients who will receive doxycycline and those who will not have comparable severity of cardiac disease, patients will be stratified according to the stage of cardiac involvement. Patients with very advanced heart dysfunction will not be enrolled in the trial, because preliminary data indicate that doxycycline is of little or no benefit in these subjects. Patients will be randomized to receive doxycycline or standard antibiotics in combination with anti-plasma cell therapy. Bortezomib-based treatment directed against plasma cells will be delivered according to each participating institutions' guidelines. Doxycycline will be administered at a dosage of 100 mg two times a day, which is usual in the treatment of bacterial diseases. Standard antibiotics will be delivered according to each participating institutions' guidelines (provided that drugs of the same class as doxycycline are not administered) in the control arm. Patients will be provided a diary to record possible adverse events and will be instructed accordingly. Patients will be evaluated at trial centers every 2 months for treatment efficacy and toxicity. In case of unsatisfactory response second-line therapy will be initiated. In the absence of unacceptable toxicity, doxycycline administration will be continued for the entire duration of follow-up (12 months).

ELIGIBILITY:
INCLUSION CRITERIA

1. Age ≥ 18.
2. Newly-diagnosed AL amyloidosis.
3. Confirmed diagnoses of AL amyloidosis by the following:

   1. histochemical diagnoses of AL amyloidosis determined by polarizing light microscopy of green birefringent material in Congo red stained issue specimens OR characteristic electron microscopy appearance AND
   2. confirmatory electron microscopy immunohistochemistry OR mass spectroscopy of AL amyloidosis. Confirmation of amyloid type can be omitted in patients with a clear-cut clinical evidence of AL amyloidosis (e.g. cardiac and renal involvement, soft tissue involvement) in the presence of a monoclonal component.
4. Cardiac involvement as defined by ALL of the following:

   1. Either an endomyocardial biopsy consistent with AL amyloidosis OR an echocardiogram demonstrating a mean left ventricular wall thickness in diastole >12 mm in the absence of other causes (e.g., severe hypertension, aortic stenosis) which would adequately explain the degree of wall thickening .
   2. Cardiac stage II disease: either cTnT > 0.035 ng/mL (or in place of cTnT the cTnI > 0.10 ng/mL or hs-cTnT >77 ng/L) or simultaneous NT-proBNP >332 ng/L OR patients with cardiac stage IIIa: both cTnT > 0.035 ng/mL (or in place of cTnT the cTnI > 0.10 ng/mL or hs-cTnT >77 ng/L) and simultaneous NT-proBNP >332 ng/L and NT-proBNP ≤8500 ng/L.
5. Planned bortezomib-based therapy.
6. Total bilirubin <1.5 × upper reference limit (url), patients with Gilbert disease who have a total bilirubin, predominantly unconjugated >1.5 × url without any other liver function test abnormalities are still eligible.
7. Alkaline phosphatase <5 × url.
8. Alanine aminotransferase <3 × url.
9. Systolic blood pressure 90-180 mmHg.
10. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 14 days prior to the first administration of study drug and perform a pregnancy test every 4 weeks to rule out pregnancy, they must agree to use highly effective physician-approved contraception 30 days prior to the first study drug administration.

    Highly-effective contraceptive methods with a Pearl Index lower than 1 are: Oral hormonal contraception ('pill') (as far as its efficacy is not expected to be impaired during the trial, e.g. with IMPs that cause vomiting and diarrhoea or interfere with hormone metabolism, adequate safety cannot be assumed), Dermal hormonal contraception (e.g. contraceptive patch), Vaginal hormonal contraception (NuvaRing®), Long-acting injectable contraceptives, Tubal ligation (female sterilisation), Double barrier methods. This means that the following are not regarded as safe: condom plus spermicide, simple barrier methods (vaginal pessaries, condom, female condoms), copper spirals, the rhythm method, basal temperature method, and the withdrawal method (coitus interruptus).

    The following duration of highly effective contraception is necessary: Bortezomib: during and until 3 months after the end of therapy, Melphalan: during and 6 months after the end of therapy, Cyclophosphamide: during and 12 months after the end of therapy
11. Males must be surgically sterile or must agree to use highly effective physician approved contraception from 30 days prior to the first study drug administration to 90 days following the last study drug administration.
12. Ability to understand and willingness to sign an informed consent form prior to initiation of any study procedures.
13. Patient was assessed to determine ineligibility for ASCT. Patients who are eligible for high-dose chemotherapy and ASCT but decline the procedure, can be enrolled in the study.

EXCLUSION CRITERIA

1. Non-AL amyloidosis.
2. Stage IIIb (NT-proBNP >8500 ng/L and cTnI >0.1 ng/mL, or cTnT >0.035 ng/mL, or hs-cTnT >77 ng/L.
3. Previous treatment for AL amyloidosis.
4. Clinically overt multiple myeloma with lytic bone lesions.
5. Symptomatic orthostatic hypotension that in the medical judgment of the Investigator would interfere with subject's ability to safely receive treatment or complete study assessments.
6. Patients with uncontrolled infection or active malignancy with the exception of adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for 5 years.
7. Known HIV positive.
8. Pregnant or nursing women.
9. Known hypersensitivity to doxycycline, bortezomib, boron, or mannitol.
10. Treatment with drugs potentially affecting doxycycline absorption.
11. Significant acute gastrointestinal symptoms.
12. Active peptic ulceration and/or esophageal reflux disease.
13. Patients with serious medical or psychiatric illness likely to interfere with participation in this clinical study.
14. Contraindication to bortezomib based therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
proportion surviving | 12 months
  proportion surviving

CONTACTS AND LOCATIONS:
Locations (8):
- Cross Cancer Insititue, University of Alberta, Edmonton, Canada
- CHU Limoges, Limoges, France
- University Hospital, Heidelberg, Germany
- Alexandra Hospital, Athens, Greece
- Fondazione IRCCS Policlinico San Matteo, Pavia, Italy
- Hospital Clinic de Barcelona, Barcelona, Spain
- Istanbul University Cerrahpasa Faculty of Medicine, Istanbul, Turkey (Türkiye)
- University College London Medical School and Royal Free Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No